CLINICAL TRIAL: NCT01295684
Title: The Influence Of Cranberry Juice On Risk Factors For Cardiovascular Disease
Brief Title: Cranberry Juice and Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Janet Novotny, Ph. D., USDA
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2010-085
Record Dates: First submitted 2010-05-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Cardiovascular Disease
Keywords: cranberry; cardiovascular; adhesion; polyphenol
MeSH Terms: conditions — Cardiovascular Diseases; Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Base diet supplemented with two 8 ounce servings of a color and flavor matched placebo beverage.
  Interventions: Other: Placebo
- Cranberry Juice (Experimental): Base diet supplemented with two 8 ounce servings of low calorie cranberry juice per day.
  Interventions: Other: Cranberry juice

INTERVENTIONS:
Other: Cranberry juice — base diet supplemented with two 8 ounce servings of low calorie cranberry juice per day
  Arms: Cranberry Juice
Other: Placebo — base diet supplemented with two 8 ounce servings of a color and flavor matched placebo beverage
  Arms: placebo

SUMMARY:
Previous studies have shown that consumption of a low calorie cranberry beverage imparts a favorable impact on HDL cholesterol, LDL oxidation, and cell adhesion molecules in men. However, these studies were not well controlled. Thus, it is important to confirm these effects in a blinded, placebo-controlled feeding study. The investigators goal is to verify the cardioprotective effects of cranberries by conducting a dietary intervention trial with healthy subjects in a controlled environment.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 65 years of age
* BMI 20 to 38 kg/m2

Exclusion Criteria:

* history of bariatric or certain other surgeries related to weight control
* kidney disease, liver disease, certain cancers, gout, hyperthyroidism, untreated or unstable hypothyroidism, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Type 2 diabetes or use of glucose-lowering medication
* Have a fasting blood sugar greater than 126 mg/dL
* LDL-cholesterol less than 130 mg/dL
* fasting triglycerides greater than 300 mg/dL
* use of cholesterol-lowering medication or supplements
* use of blood pressure-lowering medication
* smoking or use of other tobacco products (within 6 months prior to the start of the study)
* unwillingness to abstain from vitamin, mineral, and herbal supplements for 2 weeks prior to the study and during the study
* use antibiotics during the study,or for 3 weeks prior to starting the study.
* history of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* weight loss of >/= 10% of your body weight within the last 12 months or plan to initiate a weight loss program during the next 10 months
* inability to eat cranberries
* inability or unwillingness to give informed consent or communicate with study staff
* self-reported history of alcohol or substance abuse within the past 12 months and/or are currently in treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers of cardiovascular disease and polyphenol absorption | Days 1&2; Days 27&28; Days 55&56
  A blood lipid panel will include plasma total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, Apo A-1, Apo A-II, Apo B, Lpa. Inflammatory markers (IL-6, IL-10, IL-1-alpha, CRP, TNF-alpha, fibrinogen, iCAM) will be determined by ELISA. Serum will be analyzed for polyphenol concentration.

SECONDARY OUTCOMES:
Change from baseline in systolic and diastolic blood pressure | Days 1, 28, and 56
  Blood pressure will be measured using a standardized protocol at the beginning, 4-week, and 8-week time points.
Change in urine metabolomics and adhesion analysis | Days 1 & 56
  Urine (24 hour cumulative and spot)will be collected at the beginning and end of each treatment period and provided to Ocean Spray for metabolomics and adhesion analysis.
Change in fecal microbiota | Days 1 & 56
  A spot fecal sample will be collected at the beginning and end of each treatment period and provided to Ocean Spray microbiota analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Novotny, Ph. D., Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA's Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Novotny JA, Baer DJ, Khoo C, Gebauer SK, Charron CS. Cranberry juice consumption lowers markers of cardiometabolic risk, including blood pressure and circulating C-reactive protein, triglyceride, and glucose concentrations in adults. J Nutr. 2015 Jun;145(6):1185-93. doi: 10.3945/jn.114.203190. Epub 2015 Apr 22. PMID 25904733